CLINICAL TRIAL: NCT03219255
Title: Relvar 100 Ellipta Special Drug Use Investigation (COPD, Long-term)
Brief Title: RELVAR® 100 ELLIPTA® Special Drug Use Investigation (COPD, Long-term)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 205653
Record Dates: First submitted 2017-07-07; First posted 2017-07-17 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Post-marketing; Chronic obstructive pulmonary disease; Drug use investigation; RELVAR 100 ELLIPTA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects receiving RELVAR 100 ELLIPTA: Subjects with a diagnosis of COPD, for which RELVAR is indicated, who are naive to RELVAR will be included.
  Interventions: Drug: RELVAR 100 ELLIPTA

INTERVENTIONS:
Drug: RELVAR 100 ELLIPTA — RELVAR 100 ELLIPTA contains fluticasone furoate, an inhaled corticosteroid and vilanterol, an ultra-long-acting Beta-2 agonist and it is indicated for the treatment of COPD (bronchitis chronic/emphysema). Post-marketing investigation of RELVAR 100 ELLIPTA will be carried out in this analysis.

SUMMARY:
This study aims to investigate the long-term safety and efficacy of RELVAR® 100 ELLIPTA® (hereinafter referred to as "Relvar") in daily clinical practice in subjects with chronic obstructive pulmonary disease (COPD), who are naive to RELVAR. A total of 1000 subjects, from approximately 200 medical institutions, will be registered for this study and 332 of them will be considered for safety analysis. In the investigation, subject registration and data collection will be conducted using an Electronic Data Capture (EDC) system. Post-registration, the investigator will monitor the information regarding the safety and efficacy of RELVAR for one year from the start date of treatment with RELVAR. Pneumonia, systemic effects caused by corticosteroids and cardiovascular events will be considered as the priority investigation matters. At the end of observation period, the investigator will enter the obtained information into the EDC system and submit it. RELVAR 100 ELLIPTA is the registered trademark of GlaxoSmithKline (GSK) group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of COPD (bronchitis chronic/emphysema) and who are naive to RELVAR will be included.

Exclusion Criteria:

* Among subjects with concomitant asthma, subjects with experience of taking RELVAR for treatment of asthma will be excluded from the investigation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will assess and collect the information about safety and effectiveness of RELVAR in approximately 1000 subjects with COPD (bronchitis chronic/emphysema), for which RELVAR is indicated, who are naïve to RELVAR.
Sampling Method: Probability Sample
Enrollment: 1047 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs), serious adverse events (SAEs) and drug related AEs | One year from the start of RELVAR treatment
  The investigator will collect the information about all AEs (e.g., a disease, symptom, abnormal laboratory value) occurring after the start of RELVAR administration, regardless of whether or not RELVAR is related to an AE. The AEs assessed as 'related' to RELVAR will be handled as adverse drug reactions (ADRs).
Number of subjects with pneumonia, systemic effects caused by corticosteroids and cardiovascular events | One year from the start of RELVAR treatment
  Pneumonia, systemic effects such as suppression of adrenal cortical function, bone disorders, eye disorders, etc. caused by corticosteroids and cardiovascular events will be considered as priority investigation matter for this investigation and its occurrence will be monitored throughout the study period.
Efficacy rate based on global efficacy assessment | One year from the start of RELVAR treatment
  The efficacy rate is the proportion of subjects assessed as "effective." Efficacy will be globally assessed based on the courses of subjective and clinical symptoms, COPD exacerbation, changes in values for respiratory function tests, change in COPD assessment test (CAT) scores, etc. during the period between the start date of treatment and the end of the observation period.
Time to COPD exacerbation | One year from the start of RELVAR treatment
  The COPD exacerbations are episodes, which may refer to an increase in the severity of disease or its sign and symptoms. The presence or absence of exacerbation for one year before and after the start of treatment with RELVAR (or at the time of withdrawal/ termination), presence or absence of hospitalization, treatment with antimicrobial agents and/or systemic steroids and exacerbation not corresponding to the above-mentioned parameters in each exacerbation episode will be determined.
Change from Baseline in CAT score | Baseline and up to one year from the start of RELVAR treatment
  The CAT is a questionnaire designed to measure the impact of COPD on subject's life and how it changes over time. Investigator will record the information of CAT completed by subjects at the start of treatment with RELVAR, Month 3 and Year 1 or at the time of withdrawal/termination.
Change from Baseline in forced expiratory volume in 1 second (FEV1) | Baseline and up to one year from the start of RELVAR treatment
  Respiratory function test will be performed by spirometry. Information regarding presence or absence of tests, date of tests, presence or absence of short-acting Beta-2 agonists within four hours before measurement, and FEV1 at the start of treatment with RELVAR, Month 3 and Year 1 or at the time of withdrawal/termination will be collected.
Change from Baseline in forced vital capacity (FVC) | Baseline and up to one year from the start of RELVAR treatment
  Respiratory function test will be performed by spirometry. Information regarding presence or absence of tests, date of tests, presence or absence of short-acting Beta-2 agonists within four hours before measurement, and FVC at the start of treatment with RELVAR, Month 3 and Year 1 or at the time of withdrawal/termination will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa

IPD SHARING:
Plan to Share IPD: No